CLINICAL TRIAL: NCT04981340
Title: The Role of Abdominal and Pelvic Floor Retraining in Children With Dysfunctional Voiding
Brief Title: Diaphragmatic Breathing Exercises and Pelvic Floor Retraining in Children With Dysfunctional Voiding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nis (Other)
Responsible Party: Principal Investigator, Vesna Zivkovic, MD, PhD, Professor of physical and rehabilitation medicine, University of Nis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43011
Record Dates: First submitted 2021-07-12; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Dysfunctional Voiding
Keywords: dysfunctional voiding; diaphragmatic breathing; urotherapy; pelvic floor exercises; The Dysfunctional Voiding and Incontinence Scoring System

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard urotherapy + Diaphragmatic breathing exercises+ pelvic floor exercises (Experimental): Diaphragmatic breathing exercises will be demonstrated by a qualified physiotherapist. Exercises will be done in lying and sitting positions respectively. In supine, with the lower extremities supported over a pillow and hands positioned on the abdominal muscles, children will be asked to inhale the air through the nose, bulge the abdomen outwards as much as possible, hold their breath for a few seconds, and then exhale slowly through pursed lips. The same exercise will be then performed in both side-lying positions and in a sitting position in front of the mirror. Children will be instructed to watch the anterior abdominal wall movement during inspiration and to repeat the same action while seated on the toilet to initiate voiding. They will be asked to perform the diaphragmatic breathing exercises daily at home.
  Interventions: Behavioral: Diaphragmatic breathing; Behavioral: Standard urotherapy
- Standard urotherapy (Active Comparator): Standard urotherapy will start with the education of the children and their parents about the normal function of the bladder and external urinary sphincter and the nature of their voiding disorder. The importance of regular fluid intake (200 ml 5-6 times per day) and regular voiding will be explained. Special voiding and defecation diaries that a child has to fill out at home will be provided. An optimal voiding posture will be demonstrated in front of a mirror: a sitting position, with feet supported, hips abducted and abdominal muscles relaxed.
  Interventions: Behavioral: Standard urotherapy

INTERVENTIONS:
Behavioral: Diaphragmatic breathing — Same as previously described
  Arms: Standard urotherapy + Diaphragmatic breathing exercises+ pelvic floor exercises
Behavioral: Standard urotherapy — Same as previously described

SUMMARY:
According to the 2016 International Children's Continence Society standardization of terminology of lower urinary tract function in children, dysfunctional voiding (DV) is a "urodynamic entity characterized by an intermittent and/or fluctuating uroflow rate due to involuntary intermittent contractions of the striated muscle of the external urethral sphincter or pelvic floor during voiding in neurologically normal individuals" . Symptoms vary from mild daytime frequency and urgency to daytime and nighttime wetting, pelvic holding maneuvers, voiding difficulties, urinary tract infections and vesicoureteral reflux (VUR).

There are several ways of treating DV, including urotherapy, pharmacotherapy, surgery in the most severe cases, and even Botulinum toxin type A application in certain children. ''Urotherapy'' stands for non-surgical, non-pharmacologic treatment of lower urinary tract function and can be defined as a bladder re-education or rehabilitation program aiming at correction of filling and voiding difficulties. It involves the change of habits that a child has acquired during the period of toilet training and the development of motor control of the micturition reflex. Urotherapy starts with both parental and child education about the importance of regular hydratation and voiding, constipation treatment and genital hygiene. Together with this standard treatment, the pelvic floor muscle (PFM) retraining is initiated, and it includes pelvic floor exercises and various forms of biofeedback (visual, tactile, auditory, electromyography) with the same aim in mind - to help the child establish pelvic floor awareness and control, and relearn pelvic floor muscle relaxation.

During the past decade, it has been shown that the PFMs are not an isolated unit, but a part of the abdominal capsule, which they form together with the diaphragm, superficial and deep abdominal muscles. As lower abdominal and PFM act synergistically, it is important that both be relaxed during voiding. Diaphragmatic breathing exercises are easy to learn and serve to teach the children abdominal relaxation.

ELIGIBILITY:
Inclusion Criteria:

1. Proven dysfunctional voiding according to the ICCS criteria
2. Signed informed consent by parents motivated to participate in the study
3. Previous treatment by pediatricians in primary care with timed voiding, hydratation and constipation management for three months with no significant success

Exclusion Criteria:

1. Neurological disorders
2. Monosymptomatic nocturnal enuresis
3. Mental retardation
4. Structural abnormalities of the lower urinary tract -

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-18 (Estimated); Primary Completion 2022-09-29 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with cured or improved urinary incontinence, nocturnal enuresis, urinary tract infections and constipation at the end of the trial in each group of patients | 12 months
  During the treatment period, all children in both groups will be asked to keep: a 48hr daytime frequency and volume chart, and a 7-day bladder and defecation diary. Children will be re-evaluated each month after the beginning of the therapy. The analysis of the diaries and charts will start with each visit to the Clinic, noticing changes in urinary incontinence, nocturnal enuresis, defecation frequency and urinary tract infections.
Number of patients with improved uroflowmetry parameters and curve type | 12 months
  Uroflowmetry with pelvic floor electromyography and post-void residual (PVR) urine measurement will be performed in both groups during monthly visits. It will be carried out twice as a child feels the need to void. PVR urine will be detected by ultrasound less than a minute after voiding.
Number of patients with non-, partial and full response in both groups. | 12 months
  Based on the clinical manifestations and uroflowmetry parameters, treatment result will be defined as full, partial and non-response. In children in whom urinary incontinence, nocturnal enuresis and urinary tract infections disappear entirely, treatment outcome will be described as "full response"; "partial response" when wetting episodes and urinary tract infections are reduced by more than 50%, and "non-response" when urinary incontinence, nocturnal enuresis and urinary tract infections persist. In children with constipation ≥ 3 bowel movements per week, ≤ 2 episodes of fecal incontinence per month and no abdominal pain with no laxative treatment for > 1 month will be classified as "full response".

SECONDARY OUTCOMES:
Mean pre- and post-treatment Dysfunctional voiding and Incontinence Symptoms Score in children with non-, partial and full response in both groups. | 12 months
  The Dysfunctional Voiding and Incontinence Scoring System will be completed at the beginning and the end of the 12-month treatment period. This questionnaire consists of 13 questions relating to daytime and nighttime wetting, degree of wetting, frequency of urination, voiding symptoms ( straining, intermittency), pain, urgency, urge incontinence, pelvic holding maneuvers, defecation frequency, and one question concerning the impact of voiding disorder on quality of life. Parents are expected to score the frequency and intensity of wetting during the day and night in the first four questions in the presence of their child, and the last eight questions are answered in a yes or no manner. Each answer, except the last question, is scored to produce a total score of between 0 and 35. The presence of voiding dysfunction (excluding quality of life score) in both genders is indicated by a total score of 9 or more.
Number of patients with pre-treatment score ≥ 9 in children with non-/ partial and full response in both groups. | 12 months
  In order to determine sensitivity and specificity of the initial and final score in predicting treatment outcome, all children will be divided in two groups. One group will consist of all children with full response, while the second group will consist of children with partial and non-response. Individual pre- and post-treatment total scores will be compared to the treatment outcome.
Number of patients with post-treatment score < 9 in children with non-/ partial and full response in both groups. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ivona Stankovic, MD, Study Director — University of Nis Medical faculty
Locations (1):
- Medical Faculty, Niš, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695